CLINICAL TRIAL: NCT00336141
Title: Phase I/II Clinical Trial With Vorinostat and Infusional 5-FU/LV in Patients With Metastatic Colorectal Cancer Who Failed 5-FU-Based Chemotherapy
Brief Title: Vorinostat and IV Fluorouracil/Leucovorin (5FU/LV) in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3C-05-3
Record Dates: First submitted 2006-06-09; First posted 2006-06-13 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Vorinostat

ARMS (1):
- Vorinostat (Experimental)
  Interventions: Drug: Suberoylanilide hydroxamic acid

INTERVENTIONS:
Drug: Suberoylanilide hydroxamic acid — 400 mg QD (every day) for five days, followed by 9 days of no vorinostat

SUMMARY:
This protocol will investigate the use of vorinostat (suberoylanilide hydroxamic acid - SAHA) in combination with infusional 5-FU and leucovorin for the treatment of metastatic colorectal cancer patients who have failed standard 5FU regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced/metastatic colorectal cancer.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than 20 mm with conventional techniques or as > 10 mm with spiral CT scan.
* Patients must have received prior therapy (in any setting) with 5-FU, CPT-11, and oxaliplatin. Patients may have received prior erbitux and bevacizumab, but it is not required.
* Patients must have received at least one prior chemotherapy regimen for advanced disease.
* Tumor must be accessible for core biopsy at the beginning of treatment and patients have a high intratumoral TS expression level prior to the beginning of treatment.
* Age > 18 years. Because no dosing or AE data are currently available on the use of vorinostat in patients greater than 18 years of age, children are excluded from this study but will be eligible for future pediatric single-agent trials, if applicable.
* Life expectancy of > 12 weeks.
* ECOG performance status 0-2 (Karnofsky > 50%; see Appendix A).
* Patients must have normal organ and marrow function as defined below:
* leukocytes > 3,000/µL
* absolute neutrophil count > 1,500/µL
* platelets > 100,000/µL
* hemoglobin > 9 mg/dL
* total bilirubin within 1.5 x normal institutional limits
* AST (SGOT)/ALT (SGPT) greater than or equal to 2.5 X institutional upper limit of normal
* creatinine greater than or equal to 1.5 X institutional upper limit of normal OR
* creatinine clearance > 60 mL/min/1.73 m2
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of vorinostat will be determined following review by the principal investigator. (A list of medications and substances known or with the potential to interact with selected CYP450 isoenzymes is provided in Appendix B.)
* Ability to understand and the willingness to sign a written informed consent document.
* INR is ≤ 1.5 times the upper limit of normal (ULN) unless receiving therapeutic anticoagulation
* Patient is highly unlikely to conceive as indicated by at least one "yes" answer to the following questions:
* Patient is a male and agrees to use an adequate method of contraception for the duration of the study, and for 30 days after the last dose of study medication.
* Patient is a surgically sterilized female.
* Patient is a postmenopausal female ≥ 45 years of age with > 2 years since last menses.
* Patient is a non-sterilized premenopausal female and agrees to use 2 adequate barrier methods of contraception to prevent pregnancy or agrees to abstain from heterosexual activity throughout the study and for 30 days after the last dose of study medication.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from AEs due to agents administered more than 4 weeks earlier.
* Patients may not have received any other investigational agents within 28 days of study entry.
* Patients may not receive other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) while on this study.
* Patients with known brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat. These compounds include sodium butyrate, trichostatin A (TSA), trapoxin (TPX), MS-27-275 and depsipeptide.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because vorinostat is a HDAC inhibitor agent with an unknown potential for teratogenesis. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with vorinostat, breastfeeding should be discontinued before the mother is treated with study therapy.
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with vorinostat. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.
* Patient is on any systemic steroids that have not been stabilized to the equivalent of ≤ 10 mg/day prednisone during the 4 weeks prior to the start of the study drugs.
* Patient has had an acute infection requiring intravenous antibiotic, antiviral, or antifungal medications within 2 weeks prior to the start of study drugs.
* Patient has an active hepatitis B or hepatitis C infection.
* Patient has a history of GI surgery or other procedures that might, in the opinion of the investigator, interfere with the absorption or swallowing of the study drugs.
* Patient has had prescription or non-prescription drugs or other products known to influence CYP3A4 that cannot be discontinued prior to day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study medication. Refer to Appendix B for a list of commonly used moderate and potent CYP3A4 modifiers and their required washout periods.
* Patient has had prior cancer treatment with an HDAC inhibitor (e.g., Depsipeptide, MS 275, LAQ-824, PXD-101, and valproic acid). Patients who have received such agents for other indications, e.g., epilepsy, may enroll in the trial after a 30 day washout period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Toxicity | Weekly

SECONDARY OUTCOMES:
Response | Every 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States